CLINICAL TRIAL: NCT04509973
Title: Higher vs. Lower Doses of Dexamethasone in Patients With COVID-19 and Severe Hypoxia
Brief Title: Higher vs. Lower Doses of Dexamethasone for COVID-19 and Severe Hypoxia
Acronym: COVIDSTEROID2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scandinavian Critical Care Trials Group (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Centre for Research in Intensive Care (CRIC) (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Rigshospitalet, Denmark (Other); The George Institute for Global Health, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RH-ITA-009; 2020-003363-25 (EudraCT Number); 2020-07-16 (Other: Danish Medicines Agency); H-20051056 (Other: Ethic committee of the Capital Region, DK)
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Covid19; Hypoxia
Keywords: Randomised clinical trial; COVID-19; Hypoxia; Corticosteroids
MeSH Terms: conditions — COVID-19; Hypoxia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone 12 mg (Experimental): Intravenous bolus injection of dexamethasone 12 mg once daily in addition to standard care for up to 10 days. We will allow the use of betamethasone 12 mg at sites, where dexamethasone is not available.
  Interventions: Drug: Dexamethasone
- Dexamethasone 6 mg (Active Comparator): Intravenous bolus injection of dexamethasone 6 mg once daily in addition to standard care for up to 10 days. We will allow the use of betamethasone 6 mg at sites, where dexamethasone is not available.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — ATC code: H02AB02
  Other Names: Dexavit

SUMMARY:
We aim to assess the benefits and harms of higher (12 mg) vs lower doses (6 mg) of dexamethasone on patient-centered outcomes in patients with COVID-19 and severe hypoxia.

DETAILED DESCRIPTION:
Background: Preliminary results from the Randomised Evaluation of COVid-19 thERapY (RECOVERY) trial have reported a reduction in 28-day mortality with low-dose dexamethasone (6 mg) once daily versus no intervention in hospitalised patients with COVID-19; an effect that may have been more pronounced in patients with increasing hypoxia. Yet, higher doses of dexamethasone may be beneficial in patients with non-COVID-19 acute respiratory distress syndrome. At present, it is unclear what dose of dexamethasone is most beneficial in patients with COVID-19 and severe hypoxia, and clinical equipoise exists.

Objective: We aim to assess the effects of higher (12 mg) vs lower doses (6 mg) of intravenous dexamethasone on the number of days alive without life-support in adult patients with COVID-19 and severe hypoxia.

Design: International, parallel-group, centrally randomised, stratified, blinded, clinical trial.

Population: Adult patients with documented COVID-19 receiving at least 10 L/min of oxygen independent of delivery system OR mechanical ventilation.

Experimental intervention: Dexamethasone 12 mg once daily for up to 10 days in addition to standard care.

Control intervention: Dexamethasone 6 mg once daily for up to 10 days in addition to standard care.

Outcomes: The primary outcome is days alive without life support (i.e. mechanical ventilation, circulatory support, or renal replacement therapy) at day 28. Secondary outcomes are serious adverse reactions (i.e. anaphylactic reaction to hydrocortisone, new episode of septic shock, invasive fungal infection or clinically important gastrointestinal bleeding) at day 28; days alive without life support at day 90; days alive and out of hospital at day 90; all-cause mortality at day 28, 90 and 180; and health-related quality of life at day 180.

Sample size: A total of 1000 participants will be randomised in order to detect a 15% relative reduction in 28-day mortality combined with a 10% reduction in time on life support among the survivors with a power of 85%.

ELIGIBILITY:
Inclusion Criteria: All of the following must be fulfilled

* Aged 18 years or above AND
* Confirmed SARS-CoV-2 (COVID-19) requiring hospitalisation AND
* Use of one of the following:

  * Invasive mechanical ventilation OR
  * Non-invasive ventilation or continuous use of continuous positive airway pressure (CPAP) for hypoxia OR
  * Oxygen supplementation with an oxygen flow of at least 10 L/min independent of delivery system

Exclusion Criteria: We will exclude patients who fulfil any of the following criteria:

* Use of systemic corticosteroids for other indications than COVID-19 in doses higher than 6 mg dexamethasone equivalents
* Use of systemic corticosteroids for COVID-19 for 5 days consecutive days or more
* Invasive fungal infection
* Active tuberculosis
* Fertile woman (<60 years of age) with positive urine human gonadotropin (hCG) or plasma-hCG
* Known hypersensitivity to dexamethasone
* Previously randomised into the COVID STEROID 2 trial
* Informed consent not obtainable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Days alive without life support at day 28 | Day 28 after randomisation
  Days alive without life support (i.e. invasive mechanical ventilation, circulatory support or renal replacement therapy) from randomisation to day 28

SECONDARY OUTCOMES:
Number of participants with one or more serious adverse reactions | Day 28 after randomisation
  Serious adverse reactions defined as new episodes of septic shock, invasive fungal infection, clinically important gastrointestinal bleeding or anaphylactic reaction
All-cause mortality at day 28 | Day 28 after randomisation
  Death from all causes
All-cause mortality at day 90 | Day 90 after randomisation
  Death from all causes
Days alive without life support at day 90 | Day 90 after randomisation
  Days alive without life support (i.e. invasive mechanical ventilation, circulatory support or renal replacement therapy) from randomisation to day 90
Days alive and out of hospital at day 90 | Day 90 after randomisation
  Number of days alive and out of hospital not limited to the index admission
All-cause mortality at day 180 | Day 180 after randomisation
  Death from all causes
Health-related quality of life at day 180 | Day 180 after randomisation
  Assessed by EQ-5D-5L
Health-related quality of life at day 180 | Day 180 after randomisation
  Assessed by EQ-VAS

CONTACTS AND LOCATIONS:
Locations (53):
- Denmark (19):
  - Dept. of Anaesthesia and Intensive Care, Aalborg University Hospital, Denmark., Aalborg
  - Dept. of Intensive care, Aarhus University Hospital, Aarhus
  - Dept. of Intensive Care, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Dept. of Neuroanaesthesiology, Copenhagen
  - Dept. of Thoracic Anaesthesiology, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Dept of Infectious diseases, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Dept. of Intensive Care, Gentofte Hospital, Hellerup
  - Dept. of Anaesthesia and Intensive Care, Herlev Hospital, Herlev
  - Dept. of Anaesthesia, Regional Hospital West Jutland, Herning, Herning
  - Dept. of Intensive Care, Nordsjællands Hospital - Hillerød, Denmark., Hillerød
  - Hvidovre Hospital - Dept of Infectious diseases, Hvidovre
  - Hvidovre Hospital - Dept of Intensive Care, Hvidovre
  - Hvidovre Hospital - Dept of Pulmonary Medicine, Hvidovre
  - Dept. of Anaesthesia and Intensive Care, Lillebaelt Hospital, Kolding
  - Dept. of Intensive Care, Køge University Hospital, Køge
  - Dept of Intensive Care, Odense University Hospital, Odense
  - Dept. of Anaesthesia and Intensive Care, Zealand University Hospital Roskilde, Roskilde
  - Dept. of Anaesthesia, Slagelse Hospital, Slagelse
  - Dept. of Anaesthesia and Intensive Care, Viborg Hospital, Viborg
- India (16):
  - Jawahar Lal Nehru Medical Collega, AMU, Aligarh
  - Apollo Hospital, Chennai
  - Amrita Institute of Medical Sciences, Kochi
  - Bombay Hospital & Medical Research Centre, Mumbai
  - K. J. Somaiya Super Specialty Hospital, Mumbai
  - P. D. Hinduja National Hospital & Medical Research Centre, Mumbai
  - S L Raheja Fortis Hospital, Mumbai
  - Tata Memorial Hospital, Mumbai
  - Wockhardt hospitals, Mumbai
  - Indraprastha Apollo Hospital, New Delhi
  - Max Super Specialty Hospital, Saket, New Delhi
  - Symbiosis University Hospital and Research Centre, Pune
  - Vishwaraj Hospital, Pune
  - Rajendra Institute of Medical Sciences, Ranchi
  - Gotri General Hospital, Vadodara
  - Christian Medical College Vellore, Vellore
- Sweden (17):
  - Dept. of Anaesthesia and Intensive Care, Sahlgranska Universitetssjukhuset, Gothenburg
  - Dept. of Infectious Diseases, Sahlgranska Universitetssjukhuset, Gothenburg
  - Dept. of Anaesthesia and Intensive Care, Universitetssjukhuset i Linköping, Linköping
  - Dept. of Anaesthesia and Intensive Care, Skånes Universitetssjukhus (SUS) Malmö, Malmo
  - Dept. of Infectious Diseases, Skånes Universitetssjukhus (SUS) Malmö, Malmo
  - Dept. of Anaesthesia and Intensive Care, Vrinnevisjukhuset, Norrköping, Norrköping
  - Dept. of Anaesthesia and Intensive Care, Capio St Görans Sjukhus, Stockholm
  - Dept. of Anaesthesia and Intensive Care, Danderyds Sjukhuset, Stockholm
  - Dept. of Anaesthesia and Intensive Care, Karolinska Universitetssjukhuset, Huddinge, Stockholm
  - Dept. of Anaesthesia and Intensive Care, Karolinska Universitetssjukhuset, Solna, Stockholm
  - Dept. of Cardiology, Södersjukhuset, Stockholm
  - Dept. of Infectious Diseases, Danderyds Sjukhuset, Stockholm
  - Dept. of Infectious Diseases, Karolinska Universitetssjukhuset, Solna, Stockholm
  - Dept. of Infectious Diseases, Södersjukhuset, Stockholm
  - Dept. of Internal Medicine, Danderyds Sjukhuset, Stockholm
  - Dept. of Internal Medicine, Södersjukhuset, Stockholm
  - Södersjukhuset, Stockholm
- Dept. of Intensive Care Medicine, Bern University Hospital (Inselspital), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Fully de-identified IPD will be shared after the approval by the the trial management committee
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediate sharing of protocol, SAP and ICF. CSR will be shared no later than 6 months after last-patient-last-visit
Access Criteria: Contact to the trial management committee
URL: http://www.cric.nu/covid-steroid-2/

REFERENCES:
- [Derived] Granholm A, Kaas-Hansen BS, Lange T, Munch MW, Harhay MO, Zampieri FG, Perner A, Moller MH, Jensen AKG. Use of days alive without life support and similar count outcomes in randomised clinical trials - an overview and comparison of methodological choices and analysis methods. BMC Med Res Methodol. 2023 Jun 14;23(1):139. doi: 10.1186/s12874-023-01963-z. PMID 37316785
- [Derived] Granholm A, Kjaer MN, Munch MW, Myatra SN, Vijayaraghavan BKT, Cronhjort M, Wahlin RR, Jakob SM, Cioccari L, Vesterlund GK, Meyhoff TS, Helleberg M, Moller MH, Benfield T, Venkatesh B, Hammond NE, Micallef S, Bassi A, John O, Jha V, Kristiansen KT, Ulrik CS, Jorgensen VL, Smitt M, Bestle MH, Andreasen AS, Poulsen LM, Rasmussen BS, Brochner AC, Strom T, Moller A, Khan MS, Padmanaban A, Divatia JV, Saseedharan S, Borawake K, Kapadia F, Dixit S, Chawla R, Shukla U, Amin P, Chew MS, Wamberg CA, Bose N, Shah MS, Darfelt IS, Gluud C, Lange T, Perner A. Long-term outcomes of dexamethasone 12 mg versus 6 mg in patients with COVID-19 and severe hypoxaemia. Intensive Care Med. 2022 May;48(5):580-589. doi: 10.1007/s00134-022-06677-2. Epub 2022 Mar 31. PMID 35359168
- [Derived] Durr KM, Hendin A, Perry JJ. Effect of 12 mg vs 6 mg of dexamethasone on the number of days alive without life support in adults with COVID-19 and severe hypoxemia: the COVID STEROID 2 randomized trial. CJEM. 2022 Apr;24(3):266-267. doi: 10.1007/s43678-022-00293-1. Epub 2022 Mar 29. No abstract available. PMID 35349129
- [Derived] Granholm A, Munch MW, Myatra SN, Vijayaraghavan BKT, Cronhjort M, Wahlin RR, Jakob SM, Cioccari L, Kjaer MN, Vesterlund GK, Meyhoff TS, Helleberg M, Moller MH, Benfield T, Venkatesh B, Hammond NE, Micallef S, Bassi A, John O, Jha V, Kristiansen KT, Ulrik CS, Jorgensen VL, Smitt M, Bestle MH, Andreasen AS, Poulsen LM, Rasmussen BS, Brochner AC, Strom T, Moller A, Khan MS, Padmanaban A, Divatia JV, Saseedharan S, Borawake K, Kapadia F, Dixit S, Chawla R, Shukla U, Amin P, Chew MS, Wamberg CA, Gluud C, Lange T, Perner A. Dexamethasone 12 mg versus 6 mg for patients with COVID-19 and severe hypoxaemia: a pre-planned, secondary Bayesian analysis of the COVID STEROID 2 trial. Intensive Care Med. 2022 Jan;48(1):45-55. doi: 10.1007/s00134-021-06573-1. Epub 2021 Nov 10. PMID 34757439
- [Derived] COVID STEROID 2 Trial Group; Munch MW, Myatra SN, Vijayaraghavan BKT, Saseedharan S, Benfield T, Wahlin RR, Rasmussen BS, Andreasen AS, Poulsen LM, Cioccari L, Khan MS, Kapadia F, Divatia JV, Brochner AC, Bestle MH, Helleberg M, Michelsen J, Padmanaban A, Bose N, Moller A, Borawake K, Kristiansen KT, Shukla U, Chew MS, Dixit S, Ulrik CS, Amin PR, Chawla R, Wamberg CA, Shah MS, Darfelt IS, Jorgensen VL, Smitt M, Granholm A, Kjaer MN, Moller MH, Meyhoff TS, Vesterlund GK, Hammond NE, Micallef S, Bassi A, John O, Jha A, Cronhjort M, Jakob SM, Gluud C, Lange T, Kadam V, Marcussen KV, Hollenberg J, Hedman A, Nielsen H, Schjorring OL, Jensen MQ, Leistner JW, Jonassen TB, Kristensen CM, Clapp EC, Hjortso CJS, Jensen TS, Halstad LS, Bak ERB, Zaabalawi R, Metcalf-Clausen M, Abdi S, Hatley EV, Aksnes TS, Gleipner-Andersen E, Alarcon AF, Yamin G, Heymowski A, Berggren A, La Cour K, Weihe S, Pind AH, Engstrom J, Jha V, Venkatesh B, Perner A. Effect of 12 mg vs 6 mg of Dexamethasone on the Number of Days Alive Without Life Support in Adults With COVID-19 and Severe Hypoxemia: The COVID STEROID 2 Randomized Trial. JAMA. 2021 Nov 9;326(18):1807-1817. doi: 10.1001/jama.2021.18295. PMID 34673895
- [Derived] Granholm A, Munch MW, Myatra SN, Vijayaraghavan BKT, Cronhjort M, Wahlin RR, Jakob SM, Cioccari L, Kjaer MN, Vesterlund GK, Meyhoff TS, Helleberg M, Moller MH, Benfield T, Venkatesh B, Hammond N, Micallef S, Bassi A, John O, Jha V, Kristiansen KT, Ulrik CS, Jorgensen VL, Smitt M, Bestle MH, Andreasen AS, Poulsen LM, Rasmussen BS, Brochner AC, Strom T, Moller A, Khan MS, Padmanaban A, Divatia JV, Saseedharan S, Borawake K, Kapadia F, Dixit S, Chawla R, Shukla U, Amin P, Chew MS, Gluud C, Lange T, Perner A. Higher vs Lower Doses of Dexamethasone in Patients with COVID-19 and Severe Hypoxia (COVID STEROID 2) trial: Protocol for a secondary Bayesian analysis. Acta Anaesthesiol Scand. 2021 May;65(5):702-710. doi: 10.1111/aas.13793. Epub 2021 Feb 25. PMID 33583027
- See also: Trial website — http://www.cric.nu/covid-steroid-2/